CLINICAL TRIAL: NCT02695654
Title: Effectiveness of Ultrasound Guided Adductor Canal Blockade With Levobupivacaine and Clonidine on Chronic Pain in Knee Osteoarthritis
Brief Title: Effectiveness of Ultrasound Guided Adductor Canal Block on Chronic Pain in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Mensur Salihovic (Other)
Responsible Party: Sponsor-Investigator, Mensur Salihovic, Principal investigator, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Other Study IDs: KME 100/02/15
Record Dates: First submitted 2016-02-21; First posted 2016-03-01 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Levobupivacaine; Clonidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic pain in knee osteoarthritis: Ultrasound guided single shot Adductor canal block with 0,25% Levobupivacaine 14 ml and 100 mcg Clonidine
  Interventions: Drug: Levobupivacaine; Drug: Clonidine

INTERVENTIONS:
Drug: Levobupivacaine — 14 ml of 0,25 % Levobupivacaine
  Other Names: Chirocaine
Drug: Clonidine — Clonidine 100 mcg
  Other Names: Catapresan

SUMMARY:
Adductor canal block has become popular as effective mean for pain relief following knee surgery.This block has not been checked in chronic pain patients.The purpose of this study is to assess the efficacy and safety of adductor canal block on chronic knee pain in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis is serious epidemiologic problem. Knee prosthesis is successful treatment for many of patients with advanced knee osteoarthritis but there are important numbers of patients, which are not appropriate candidates for such surgery treatment. For them ,any treatment which could relieve pain in their knee would have good impact on quality of life. Adductor canal block is successfully used for relieving postoperative pain after knee surgery. Official approval from ethics committee of Republic Slovenia was obtained for this study. After being informed about the study and potential risks, all patients giving written informed consent will undergo an orthopedic examination and those with confirmed diagnosis of knee osteoarthritis lasted more than 6 months will be included in the study. Prior to start they filled Knee injury and osteoarthritis outcome(KOOS) form and estimate maximal and minimal intensity of pain in the knee .They repeat self assessment of pain at the same manner using 11 point numeric rating score(NRS) 1 week and 1 month after blockade.Measurement of maximum voluntary isometric contraction of quadriceps muscle (MVIC) ,time up and go test(TUG) and 30s chair stand test are performed by physiotherapist before block of adductor canal on the ipsilateral leg ,1 hour,1 week and 1 month after block..Block of adductor canal is performed by the same and trained anesthesiologist at the proximal part of the leg using 14 ml of Levobupivacaine and 100 mcg Clonidine mixed in the same syringe.At the conclusion of study patients filled the Knee injury and osteoarthritis outcome(KOOS) form once again.

ELIGIBILITY:
Inclusion Criteria:

Outpatients Had pain in knee at least 6 months before the study Knee osteoarthritis chronic pain was diagnosed based on medical history, knee X- ray and orthopedic examination.

A sufficient level of education to understand study procedures and be able to communicate with site personnel

-

Exclusion Criteria:

* Any cardiovascular, hepatic, or renal conditions that would compromise participation, in the opinion of the investigator
* Severe neurologic conditions interfere with knee condition
* Narcotic dependent (opioid intake more than 3 months and more than 30 mg of daily oral morphine equivalents)
* Coexisting severe hematological disorder or with deranged coagulation parameters
* Psychiatric illnesses
* Allergy to any of the drugs used in the study
* Infection or malignancy at the site of block
* Any active systemic infection

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients included in our study were sent by family physicians to our Pain ambulance and all have alredy diagnosed knee osteoarthritis chronic pain.Diagnosis was confirmed(or not) from Ortopedist engaged in our study.Estimation of appropriatness was made by anesthesiologyst.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Maximal and minimal Pain on the 11-point Numeric rating score Pain Scale (NRS -11) | Baseline ,1 hour,1 week and 4 weeks
  Numeric 11-point rating score is widely accepted self-reported score for measurement of chronic and acute pain in researches.Possible scores range are between 0-free of pain and 10-the worst imaginable pain

SECONDARY OUTCOMES:
The Knee injury and osteoarthritis outcome(KOOS) score change in percentage from baseline and 1 month following adductor canal block | Baseline and 1 month following adductor canal block
  KOOS is valid,reliable outcome measure in patients with knee osteoarthritis. usually used following knee surgery.This method is recognised as useful also in other and nonsurgical knee treatment.Shortened version widely used in North America is western Ontario and McMaster Universities Index(WOMAC)
Maximum voluntary isometric contraction of quadriceps muscle (MVIC) | prior, 1 hour ,1 week and 1 month after block measured by handheld dynamometer
  This method is used to check impact of block on contraction of quadriceps muscle.
Timed up to go test(TUG) | prior, 1 hour ,1 week and 1 month after block
  Time that patient need to stand up from a standard height armchair,walk 3 meters,go back to the chair and takes a seat.Used to assess a patients balance,risk of falling and global mobility
Satisfaction of patient | 1 month after block
  We determine whether the patient is satisfied with the result of treatment by asking the following question: "what is the least amount of success that the treatment would have to achieve by the end of the study and/or treatment for the patient to conclude that the treatment was worth it and the patient is satisfied?"
  The patient is asked to describe the minimum goal to be satisfied with the treatment in her own words, such as: "50% reduction in pain, to go to the store without assistance, to use only one cane, to not wake up with pain, to perform regular housekeeping duties at home with minimal breaks, to walk a certain distance, or to play tennis".
  At the end of the study the patient indicates whether that goal was achieved with a "yes" or "no" answer

CONTACTS AND LOCATIONS:
Overall Officials: Mensur Salihovic, Principal Investigator — University Medical Centre
Locations (1):
- University Medical Centre, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided